CLINICAL TRIAL: NCT04148456
Title: Covered Endovascular Reconstruction of Aortic Bifurcation (CERAB) Technique for Extensive Aortoiliac Occlusive Disease
Brief Title: CERAB Technique for Aortoiliac Occlusive Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Omar Mohamed Abd Elhakam Abd Elbaqi, Principal Investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CERAB for AIOD
Record Dates: First submitted 2019-10-30; First posted 2019-11-01 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2020-07

CONDITIONS: Aortoiliac Occlusive Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Aortoiliac occlusive disease (Other): This study will be carried out on patients with extensive Aortoiliac occlusive disease using the CERAB technique.
  Interventions: Procedure: Covered Endovacular Reconstruction of Aortic Bifurcation

INTERVENTIONS:
Procedure: Covered Endovacular Reconstruction of Aortic Bifurcation — * The occlusive lesion is then passed, either subintimal or endoluminal, using crossing wires and catheters.
  * After gaining re-entry into the lumen of the aorta, angiography will be confirmed proper positioning for those with a subintimal passage.
  * A 10-12 mm V12 LD balloon expandable ePTFE covered stent (Atrium Medical, Maquet Getinge Group, Hudson, NH) will be expanded in the distal aorta approximately 20 mm above the bifurcation through the 9 Fr sheath.
  * The proximal 2/3 part of the aortic stent will be flared with a larger balloon, usually 16 mm, thereby creating a funnel shaped covered stent. Subsequently, two 8 mm V12 balloon expandable ePTFE covered stents (Atrium Medical, Maquet Getinge Group, Hudson, NH) will be placed proximally in the distal 1/3 of the aortic stent, and then simultaneously deployed distally into the common iliac arteries creating a tight connection with the first aortic stent, thereby creating the new aortic bifurcation.

SUMMARY:
To evaluate the safety and efficacy of the CERAB technique as an alternative to surgical reconstruction for treatment of aorto-iliac occlusive disease.

DETAILED DESCRIPTION:
According to the Trans-Atlantic Inter-society Consensus (TASC-II), bypass grafting is the treatment of choice for extensive aortoiliac occlusive disease (AIOD) due to the good long-term patency rates. However, surgical reconstruction is associated with peri-operative morbidity and mortality.

Kissing stent technique was introduced as an endovascular treatment alternative for bilateral aortoiliac occlusive disease in 1991. Reported technical success rates varied with the use of bare metal stents in extensive AOID.

The COBEST trial showed that covered balloon expandable stents (CBES) have a superior primary patency rate and clinical improvement outcome at 24 months when compared with bare metal stents. CBES may immediately reduce the risk of procedural complications such as dissection, perforation, in-stent stenosis, and embolization.

In 2013, CERAB technique was introduced to improve endovascular treatment results by a more anatomical and physiological reconstruction, with a subsequent better clinical outcome.

The CERAB technique was developed to overcome the anatomical and physiological disadvantages of kissing stents such as flow disturbances leading to turbulence and stasis of blood, which may cause thrombus formation and intimal neohyperplasia.

The early results of the CERAB configuration are promising at 1-year follow up in a group of 130 patients with AOID and the 30-day major complication rate was 7.7%.

CERAB and Chimney CERAB (C-CERAB) techniques may change the treatment algorithm of AIOD and juxta-renal occlusive disease. It appears to be a safe and feasible alternative with promising results, being a valid alternative for surgery and/or kissing stents.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 years and older patients.
2. Patient presented with disabling claudication pain.
3. Patient presented with rest pain.
4. Patient presented with gangrene or atrophic changes.
5. Provided written informed consent.
6. Eligible anatomy for CERAB technique.
7. TASC- (II) classification as assigned in the study protocol (specified type B, C and D lesions).

Exclusion Criteria:

1. Age less than 18 years old.
2. Patients with acute limb ischemia.
3. Patients treated with open surgery and other endovascular techniques such as kissing stenting.
4. CERAB configuration extending into aneurysmatic infrarenal aorta.
5. Patient's life expectancy <2 years as judged by the investigator.
6. Patient has a psychiatric or other condition that may interfere with the study.
7. Patient has a known allergy to any device component.
8. Patients with a systemic infection who may be at increased risk of endovascular graft infection.
9. Patient has a coagulopathy or uncontrolled bleeding disorder.
10. Patient had a recent cerebrovascular accident (CVA) or a myocardial infarction (MI) within the prior three months.
11. Patient is pregnant (Female patients of childbearing potential only).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Primary patency | 12 months
  uninterrupted patency in the absence of re-stenosis or occlusion, without any procedures performed on the vessel or stent.
Technical success | 1 month
  successful implantation of the CERAB device restoring blood flow with <30% residual stenosis without conversion to open repair during the 30-days after implantation

SECONDARY OUTCOMES:
Secondary patency | 12 months
  patency achieved by all procedures aimed at recanalizing an occluded CBES, thereby preserving the endograft.
Freedom from target lesion revascularization (TLR) | 12 months
  an open endograft without procedures performed for re-stenosis or occlusion leading to symptoms requiring an intervention.
Clinical improvement | 12 months
  hemodynamic improvement with an increase of at least 0.10 in ABI, combined with a symptomatic improvement of at least one Rutherford category.
Re-stenosis | 12 months
  a lesion with a peak systolic value (PSV) ratio >2.5 as measured in the endograft and proximal or distal to the endograft or an angiographic diameter reduction of >50%.
Limb salvage rate | 12 months
  all patients without above ankle amputations
Minor complications | 12 months
  those that were only temporary leading to impairment, whereas major complications were defined by permanent damage or death.

CONTACTS AND LOCATIONS:
Overall Officials: omar M Abd Elhakam, Doctor, Principal Investigator — Assiut University; Ayman E Hassaballah, Professor, Study Director — Assiut University; Haitham A Hassan, Doctor, Study Chair — Assiut University; Ahmed K Sayed, Doctor, Study Chair — Assiut University

REFERENCES:
- [Background] Norgren L, Hiatt WR, Dormandy JA, Nehler MR, Harris KA, Fowkes FG; TASC II Working Group. Inter-Society Consensus for the Management of Peripheral Arterial Disease (TASC II). J Vasc Surg. 2007 Jan;45 Suppl S:S5-67. doi: 10.1016/j.jvs.2006.12.037. No abstract available. PMID 17223489
- [Background] Kuffer G, Spengel F, Steckmeier B. Percutaneous reconstruction of the aortic bifurcation with Palmaz stents: case report. Cardiovasc Intervent Radiol. 1991 May-Jun;14(3):170-2. doi: 10.1007/BF02577722. No abstract available. PMID 1878908
- [Background] Grimme FA, Goverde PA, Van Oostayen JA, Zeebregts CJ, Reijnen MM. Covered stents for aortoiliac reconstruction of chronic occlusive lesions. J Cardiovasc Surg (Torino). 2012 Jun;53(3):279-89. PMID 22695260
- [Background] Bosiers M, Iyer V, Deloose K, Verbist J, Peeters P. Flemish experience using the Advanta V12 stent-graft for the treatment of iliac artery occlusive disease. J Cardiovasc Surg (Torino). 2007 Feb;48(1):7-12. PMID 17308516
- [Background] Grimme FA, Spithoven JH, Zeebregts CJ, Scharn DM, Reijnen MM. Midterm outcome of balloon-expandable polytetrafluoroethylene-covered stents in the treatment of iliac artery chronic occlusive disease. J Endovasc Ther. 2012 Dec;19(6):797-804. doi: 10.1583/JEVT-12-3941MR.1. PMID 23210879
- [Background] Grimme FA, Reijnen MM, Pfister K, Martens JM, Kasprzak P. Polytetrafluoroethylene covered stent placement for focal occlusive disease of the infrarenal aorta. Eur J Vasc Endovasc Surg. 2014 Nov;48(5):545-50. doi: 10.1016/j.ejvs.2014.08.009. Epub 2014 Sep 11. PMID 25218651
- [Background] Sabri SS, Choudhri A, Orgera G, Arslan B, Turba UC, Harthun NL, Hagspiel KD, Matsumoto AH, Angle JF. Outcomes of covered kissing stent placement compared with bare metal stent placement in the treatment of atherosclerotic occlusive disease at the aortic bifurcation. J Vasc Interv Radiol. 2010 Jul;21(7):995-1003. doi: 10.1016/j.jvir.2010.02.032. Epub 2010 Jun 11. PMID 20538478
- [Background] Palmaz JC, Encarnacion CE, Garcia OJ, Schatz RA, Rivera FJ, Laborde JC, Dougherty SP. Aortic bifurcation stenosis: treatment with intravascular stents. J Vasc Interv Radiol. 1991 Aug;2(3):319-23. doi: 10.1016/s1051-0443(91)72250-1. PMID 1839237
- [Background] Mwipatayi BP, Thomas S, Wong J, Temple SE, Vijayan V, Jackson M, Burrows SA; Covered Versus Balloon Expandable Stent Trial (COBEST) Co-investigators. A comparison of covered vs bare expandable stents for the treatment of aortoiliac occlusive disease. J Vasc Surg. 2011 Dec;54(6):1561-70. doi: 10.1016/j.jvs.2011.06.097. Epub 2011 Sep 9. PMID 21906903
- [Background] Goverde PC, Grimme FA, Verbruggen PJ, Reijnen MM. Covered endovascular reconstruction of aortic bifurcation (CERAB) technique: a new approach in treating extensive aortoiliac occlusive disease. J Cardiovasc Surg (Torino). 2013 Jun;54(3):383-7. PMID 23640357
- [Background] Saker MB, Oppat WF, Kent SA, Ryu RK, Chrisman HB, Nemcek AA, Pearce W, Pearce W, Vogelzang R. Early failure of aortoiliac kissing stents: histopathologic correlation. J Vasc Interv Radiol. 2000 Mar;11(3):333-6. doi: 10.1016/s1051-0443(07)61426-2. No abstract available. PMID 10735428
- [Background] Taeymans K, Goverde P, Lauwers K, Verbruggen P. The CERAB technique: tips, tricks and results. J Cardiovasc Surg (Torino). 2016 Jun;57(3):343-9. Epub 2016 Mar 24. PMID 27012930
- [Background] Groot Jebbink E, Grimme FA, Goverde PC, van Oostayen JA, Slump CH, Reijnen MM. Geometrical consequences of kissing stents and the Covered Endovascular Reconstruction of the Aortic Bifurcation configuration in an in vitro model for endovascular reconstruction of aortic bifurcation. J Vasc Surg. 2015 May;61(5):1306-11. doi: 10.1016/j.jvs.2013.12.026. Epub 2014 Jan 29. PMID 24486037
- [Background] Grimme FA, Goverde PC, Verbruggen PJ, Zeebregts CJ, Reijnen MM. Editor's Choice--First Results of the Covered Endovascular Reconstruction of the Aortic Bifurcation (CERAB) Technique for Aortoiliac Occlusive Disease. Eur J Vasc Endovasc Surg. 2015 Nov;50(5):638-47. doi: 10.1016/j.ejvs.2015.06.112. Epub 2015 Sep 3. PMID 26343310
- [Background] Rutherford RB, Baker JD, Ernst C, Johnston KW, Porter JM, Ahn S, Jones DN. Recommended standards for reports dealing with lower extremity ischemia: revised version. J Vasc Surg. 1997 Sep;26(3):517-38. doi: 10.1016/s0741-5214(97)70045-4. PMID 9308598